CLINICAL TRIAL: NCT04473183
Title: Epidemiologic Assessment of SARS-CoV-2 Prevalence in Minnesota
Brief Title: Epidemiologic Assessment of SARS-CoV-2 (COVID-19) Prevalence in Minnesota
Status: Withdrawn | Type: Observational
Why Stopped: PI left the University, and the study was not funded.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: SURG-2020-28863
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Covid19; SARS-CoV Infection; SARS-CoV-2; Corona Virus Infection
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Coronavirus Infections | interventions — Specimen Handling; Fertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — With the participant's approval, and as approved by IRB, de-identified biological samples will be stored and tested for anti- SARS-CoV-2 IgG and IgM. These samples may be used in future COVID-19 studies to develop assays or study other features of the disease. These leftovers may be used for multiple basic science analysis and potentially for genetic testing. The consent process will explain this to prospective participants.
  During the conduct of the study, an individual participant can choose to withdraw consent to have biological specimens stored for future research. However, withdrawal of consent with regard to biosample storage will not be possible after the study is completed. The consent process will explain this to prospective participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General Healthy Population: Participants in this group are part of the general healthy population of adults 18 years-of-age and older, not known to be exposed to the virus as reported by potential participants and who have not sought medical help in the previous 4 months.
  Interventions: Diagnostic Test: Specimen Collection; Diagnostic Test: Surveys
- Medical School Residents: Participants in this group are medical school residents.
  Interventions: Diagnostic Test: Specimen Collection; Diagnostic Test: Surveys
- Individuals who are HIV positive: Participants in this group are HIV positive.
  Interventions: Diagnostic Test: Specimen Collection; Diagnostic Test: Surveys

INTERVENTIONS:
Diagnostic Test: Specimen Collection — Blood: Two tubes of blood (up to 10 ml each) will be drawn from participants and will be collected by experienced phlebotomists.
  Nasal, oral, and rectal swabs: Nasal, oral, and rectal swabs are optional specimens that patients may be asked to donate. If prospective consent is provided, swabs will be self-collected by participants after receiving clear instructions from the team and collected in the dedicated container.
  Saliva: Saliva is an optional specimen that patients may be asked to donate. If prospective consent is provided, whole saliva samples will be self-collected by participants using a pad placed between the cheek and gum for 2-5 minutes or collecting the saliva directly to a sterile container.
Diagnostic Test: Surveys — Participants will be asked to fill out a brief online survey that will investigate symptoms consistent with SARS-CoV-2 infection in the past 3 months and the geographic location of the clinic(s) they work in (if a resident of a medical school) and their comorbidities related to SARS-CoV-2.

SUMMARY:
The purpose of this epidemiologic study is to estimate the prevalence and incidence of anti-SARS-CoV-2 antibodies in at-risk, exposed, affected populations. The study will also estimate the risk of SARS-CoV-2 exposure in target population.

DETAILED DESCRIPTION:
This study is not for real-time diagnostic purposes, guidance for patient care, or the development of a diagnostic test. The research tests performed for this study will not be prioritized over clinical care samples, that research samples will be batched and tested after clinical care samples. This study is a population-based epidemiologic analysis of prevalence of various groups of persons.

Group (1) general healthy population. People 18 years of age and older that have not tested positive for SARS-CoV-2 and who have not sought medical help in the previous 4 months.

Group (2) Medical School Residents , 18 years of age and older that have not tested positive for SARS-CoV-2 Group (3) Individuals who are HIV positive. People 18 years of age and older that have not tested positive for SARS-CoV-2

ELIGIBILITY:
Inclusion Criteria:

* Participants in Group 1 (General Healthy Population) must have no known exposure to SARS-CoV-2 and have not sought medical help in the previous 4 months for SARS-CoV-2-related symptoms
* Participants in Group 2 must be currently enrolled in a medical residency program
* Participants in Group 3 must currently test positive for HIV infection

Exclusion Criteria:

* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the participant or the quality of the data (e.g., someone not able to answer the questionnaire because of a psychological condition or an anxiety disorder that is severe).
* Contraindication for routine blood draws (e.g., severe anemia, hemophilia, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 are members of general healthy population. Group 2 are medical residents. Group 3 are individuals who test positive for HIV infection.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-07-21 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Symptomatic Infection | 1 year
  Prevalence of symptomatic infection will be reported as the percent of participants in each group who test positive for SARS-CoV-2 infection and self-report symptoms of SARS-CoV-2 infection.
Prevalence of Subclinical Infection | 1 year
  Prevalence of subclinical infection will be reported as the percent of participants in each group who test positive for SARS-CoV-2 infection and self-report no symptoms of SARS-CoV-2 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Schifanella, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided